CLINICAL TRIAL: NCT00091169
Title: Phase III Randomized Placebo-Controlled Trial to Determine Efficacy of Levocarnitine for Fatigue in Patients With Cancer
Brief Title: Levocarnitine in Treating Fatigue in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: E4Z02; E4Z02 (Other: Eastern Cooperative Oncology Group); U10CA023318 (NIH); CDR0000384087 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: fatigue; unspecified adult solid tumor, protocol specific; levocarnitine; depression; pain; carnitine deficiency
MeSH Terms: conditions — Fatigue; Depression; Pain; Systemic carnitine deficiency | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive oral levocarnitine (L-carnitine) twice daily on weeks 1-4.
  Interventions: Dietary Supplement: levocarnitine
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily on weeks 1-4.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: levocarnitine — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Levocarnitine may help improve energy levels in cancer patients.

PURPOSE: This randomized phase III trial is studying how well levocarnitine works compared to a placebo in treating fatigue in cancer patients.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

* Compare the efficacy of levocarnitine (L-carnitine) supplementation vs placebo for the management of fatigue in patients with cancer.

Secondary Objectives:

* Assess the effect of levocarnitine on pain, depression and performance status at 4 and 8 weeks of follow-up.
* Determine the prevalence of serum carnitine deficiency in patients treated with these regimens.
* Explore the association between carnitine deficiency and fatigue.
* Present the toxicity profiles of all patients.

Correlative Objective:

* Measure serum levels of the pro-inflammatory cytokines and growth factors and correlate with fatigue and other onco-behavioral symptoms.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to gender, ECOG performance status (0-1 vs 2-3), and concurrent chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms in a 1:1 ratio.

* Arm I (levocarnitine): Patients receive oral levocarnitine (L-carnitine) twice daily (2000 mg/day) on weeks 1-4.
* Arm II (placebo): Patients receive oral placebo twice daily (2000 mg/day) on weeks 1-4.

The dose was titrated over a 2-day period (i.e. two 500 mg doses the first day and two 1000 mg doses the second day) to avoid gastrointestinal side effects. Patients then continued to receive two daily doses of 1000 mg on days 3 to 28.

After week 4, all patients (on both arms) receive open-label oral L-carnitine twice daily on weeks 5-8 (extension phase) administered in the same fashion as during the first 4 weeks. For patients who had received a dose modification during weeks 1 to 4, they received the same reduced dose during the extension phase (without titration)

Fatigue, pain, and depression are assessed at baseline and then at weeks 4 and 8.

PROJECTED ACCRUAL: A total of 352 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an invasive malignant disorder
* Moderate to severe fatigue within the past 4 weeks, defined as a score of ≥ 2 (on a scale of 0-4) on the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) question "I feel fatigued"
* Age 18 and over
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-3
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

Exclusion Criteria:

* Brain metastases
* Hemoglobin < 9 g/dL, taken <=4 weeks prior to registration
* Severe, uncontrolled liver disease
* Evidence of severely compromised renal function including any 1 of the following:

  * Renal failure
  * End stage renal disease
  * Ongoing renal dialysis
* Severe, uncontrolled cardiovascular disease
* Severe, uncontrolled pulmonary disease
* Pregnant or nursing
* History of seizures
* Known sensitivity to carnitine
* Delirium
* Nausea > grade 1
* Taking any form of levocarnitine (L-carnitine) supplementation or nutritional supplements containing carnitine within 2 months prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2005-12-16 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Cruciani, MD, PhD, Study Chair — Beth Israel Medical Center - Petrie Division; Russell K. Portenoy, MD, Study Chair — Beth Israel Medical Center - Petrie Division
Locations (116):
- United States (116):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Lynn Regional Cancer Center at Boca Raton Community Hospital - Main Center, Boca Raton, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Beth Israel Medical Center - Petrie Division, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Cruciani RA, Zhang JJ, Manola J, Cella D, Ansari B, Fisch MJ. L-carnitine supplementation for the management of fatigue in patients with cancer: an eastern cooperative oncology group phase III, randomized, double-blind, placebo-controlled trial. J Clin Oncol. 2012 Nov 1;30(31):3864-9. doi: 10.1200/JCO.2011.40.2180. Epub 2012 Sep 17. PMID 22987089
- [Result] Rich TA, Manola J, Cella D, et al.: An evaluation of serum cytokine levels and fatigue and depression in ECOG E4Z02. [Abstract] J Clin Oncol 29 (Suppl 15): A-9046, 2011.
- [Result] Rich TA, Fisch MJ, Manola J, et al.: Analysis of cytokines in ECOG E4Z02: A phase III randomized study of l-carnitine supplementation for fatigue in patients with cancer. [Abstract] J Clin Oncol 27 (Suppl 15): A-9635, 2009.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on 11/3/2005, accrued its first patient 12/16/2005, suspended on 5/4/2006 after reaching its original accrual goal (160 eligible patients), reactivated on 9/6/2006 after the accrual target amendment (286 eligible patients) was approved, and closed on 1/23/2007 with a total accrual of 376 patients.
Groups:
- Levocarnitine: Patients receive oral levocarnitine (L-carnitine) twice daily on weeks 1-4.
  levocarnitine: Given orally
- Placebo: Patients receive oral placebo twice daily on weeks 1-4.
  placebo: Given orally
Period: Overall Study
Arm/Group | Levocarnitine | Placebo
Started | 189 | 187
Treated | 163 | 170
Completed | 132 | 134
Not Completed | 57 | 53
Not completed — Disease progression | 3 | 1
Not completed — Adverse Event | 11 | 17
Not completed — Death | 4 | 1
Not completed — Withdrawal by Subject | 10 | 13
Not completed — Other | 3 | 4
Not completed — Not start protocol therapy | 26 | 17

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Levocarnitine | Placebo | Total
Number analyzed (Participants) | 189 | 187 | 376
Age, Continuous [Median (Full Range); unit: years] | 64 [29 to 91] | 62 [30 to 88] | 63 [29 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 79 | 190
  Male | 78 | 108 | 186

OUTCOME MEASURES:

1. Primary Outcome: Mean Score Change in Fatigue Measured With Brief Fatigue Inventory From Baseline to 4 Weeks
Description: Fatigue was measured using Brief Fatigue Inventory (BFI). The average of all 9 items included in the scale (range: 0-10) was used to measure fatigue level, and a higher average represented worse fatigue. Score change= BFI score at 4 weeks - BFI score at baseline.
Time Frame: assessed at baseline and 4 weeks after randomization
Population: All randomized patients
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Levocarnitine | Placebo
Number analyzed (Participants) | 189 | 187
units on a scale | -0.96 [-1.32 to -0.60] | -1.11 [-1.44 to -0.78]
Statistical Analysis 1: Comparison: Levocarnitine vs Placebo; Test type: Superiority or Other; p = 0.57, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Mean Score Change in Fatigue Measured With FACIT-F From Baseline to 4 Weeks
Description: Fatigue was measured using Functional Assessment of Cancer Therapy- Fatigue subscale (FACIT-F). The sum of the scores for all 13 items (range: 0-52) included in the scale was used to measure fatigue level, and lower score represented worse fatigue. Score change= FACIT-F score at 4 weeks - FACIT-F score at baseline.
Time Frame: assessed at baseline and 4 weeks after randomization
Population: All randomized patients who reported FACIT-F score at both baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Levocarnitine | Placebo
Number analyzed (Participants) | 145 | 139
units on a scale | 5.36 [3.71 to 7.01] | 4.04 [2.39 to 5.69]
Statistical Analysis 1: Comparison: Levocarnitine vs Placebo; Test type: Superiority or Other; p = 0.64, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Mean Score Change in Depression Measured With CES-D Between 4 Weeks and Baseline
Description: Depression was measured using Center for Epidemiologic Studies Depression Scale (CES-D). The sum of the scores for all 20 items (range: 0-60) was used to assess depression level, and higher scores indicated a higher level of depression. Score change= CES-D score at 4 weeks - CES-D score at baseline.
Time Frame: assessed at baseline and 4 weeks after randomization
Population: All randomized patients who reported CES-D score at both baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Levocarnitine | Placebo
Number analyzed (Participants) | 145 | 139
units on a scale | -3.05 [-4.45 to -1.65] | -2.91 [-4.21 to -1.61]
Statistical Analysis 1: Comparison: Levocarnitine vs Placebo; Test type: Superiority or Other; p = 0.93, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mean Score Change in Pain Measured With Brief Pain Inventory From Baseline to 4 Weeks
Description: Pain was measured using Brief Pain Inventory (BPI). The mean of the 4 severity items (range: 0-10 with 0 representing no pain and 10 representing pain as bad as you can imagine) was used to measure pain severity. Score change= BPI score at 4 weeks - BPI score at baseline.
Time Frame: assessed at baseline and 4 weeks after randomization
Population: All randomized patients who reported BPI score at both baseline and 4 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Levocarnitine | Placebo
Number analyzed (Participants) | 133 | 138
units on a scale | -0.19 [-0.525 to 0.145] | -0.08 [-0.434 to 0.274]
Statistical Analysis 1: Comparison: Levocarnitine vs Placebo; Test type: Superiority or Other; p = 0.61, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Prevalence of Carnitine Deficiency at 4 Weeks
Description: Carnitine deficiency is defined as a ratio of acylcarnitine (total-free) to free carnitine > 0.4 μmol/L or free carnitine < 35 μmol/L for males and < 25 μmol/L for females.
Time Frame: assessed at 4 weeks after randomization
Population: All randomized patients who had carnitine data at 4 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 133 | 132
proportion of participants | 0.113 [0.064 to 0.179] | 0.333 [0.254 to 0.421]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority or Other; p = 0.00001, Fisher Exact

6. Secondary Outcome: Proportion of Patients With Stable or Improving Performance Status at 4 Weeks
Description: Performance status (PS) was measured using Eastern Cooperative Oncology Group performance status scale. Lower score represents better PS. Change in PS was calculated by PS at week 4- PS at baseline. Patients with negative value for change in PS were considered to have stable or improving PS.
Time Frame: assessed at baseline and 4 weeks after randomization
Population: All randomized patients who had performance status data at baseline and 4 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 155 | 160
proportion of participants | 0.806 [0.735 to 0.865] | 0.875 [0.814 to 0.922]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority or Other; p = 0.677, Fisher Exact

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Levocarnitine | Placebo
Serious Adverse Events (participants affected / at risk) | 8/166 | 8/171
Other Adverse Events (participants affected / at risk) | 10/166 | 9/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levocarnitine (N=166) | Placebo (N=171)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Platelets decreased (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Death - disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levocarnitine (N=166) | Placebo (N=171)
Anemia (Blood and lymphatic system disorders) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less